CLINICAL TRIAL: NCT04198181
Title: Clinical Evaluation of the Effectiveness and Safety of Resective Epilepsy Surgery for Tuberous Sclerosis Complex Related Epilepsy
Brief Title: The Effectiveness and Safety of Resective Epilepsy Surgery for TRE
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Shenzhen Children's Hospital (Other Government); Tiantan Hospital, Capital Medical University (Unknown); Peking University People's Hospital (Other); Guangdong 999 Brain Hospital (Other); Xinqiao Hospital, Amry Medical University (Unknown); Shandong Provincial Hospital (Other Government); West China Hospital (Other); Henan Provincial People's Hospital (Other); Shanghai Children's Hospital (Other); First Medical Center, PLA General Hospital (Unknown); Fourth Medical Center, PLA General Hospital (Unknown); The First Affiliated Hospital of University of Science and Technology of China (Other); Ruijin Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Xuanwu Hospital, Beijing (Other); The First Hospital of Jilin University (Other); Xiangya Hospital of Central South University (Other); Beijing Sanbo Brain Hospital (Other); Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shuli Liang, Director of Functional Neurosurgery, Beijing Children's Hospital
Other Study IDs: TRE-RES
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-05

CONDITIONS: Tuberous Sclerosis Complex; Epilepsy
Keywords: epilepsy; tuberous sclerosis complex; resective epilepsy surgery
MeSH Terms: conditions — Tuberous Sclerosis; Epilepsy | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Patients in the surgery group will accept exclusive rational medicine therapy.
- Surgery Group: Patients in the surgery group will undergo resective surgery combined with rational medicine therapy.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Resective surgery included lobectomy (partial or total brain lobe resection), tuberectomy (epileptogenic tuber resection), and tuberectomy plus (resection of epileptogenic tuber and perituberal gyri). Tuberectomy was typically performed on the epileptogenic tuber within or near an eloquent area. Lobectomy was performed in patients with large epileptogenic tubers in the brain lobes. Multiple lobectomies, tuberectomies, tuberectomies plus, and lobectomy combined with tuberectomy/tuberectomies plus were further performed in patients with multiple epileptogenic tubers.
  Groups: Surgery Group

SUMMARY:
A prospective cohort studies to identify clinical seizure control, cognitive changes, and safety in resective epilepsy surgery in patients with TSC-related drug-resistant epilepsy.

DETAILED DESCRIPTION:
Two hundred candidates are recruited and assigned to the control and surgery groups with 100 cases in each group, respectively. All patients will accept first-stage pre-enrollment evaluations and patients in surgery group will accept second-stage invasive evaluation.

All patients will be advised to visit the hospitals for examination each year after enrollment. Seizure outcomes will be assessed with reference to patients' seizure diaries and caregivers' oral statements by both neurosurgeons and neurologists.

All adverse effects will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 (2017).

Statistical analyses were conducted using SPSS (version 26.0, IBM, USA), Stata (version 16.0, Stata Corp LLC, USA), and R (version 4.3.3, R Foundation for Statistical Computing, Austria). Outcomes were presented according to data type as percentages, mean ± standard deviation, or median (interquartile range, IQR).

Multiple imputation was employed to address missing data for IQ and QOL at enrollment and the 2-year follow-up. A sensitivity analysis was conducted to assess the robustness of the multiple imputation results. The "mi impute regress" statement in Stata facilitated the multiple imputations. 20 T-tests were utilized for comparing continuous variables, with results reported as mean ± standard deviation. The Mann-Whitney U test was applied for non-normally distributed continuous variables, presenting results as median values and IQRs. Chi-square and Fisher's exact tests were used for univariate analyses. A significance level of p < 0.05 was established.

To account for differences in covariates between the surgery and medicine groups, propensity score matching (PSM) was performed. Based on PSM, Kaplan-Meier curves and the log-rank test were utilized to analyze time-to-seizure recurrence differences between the surgery and medicine groups. Additionally, multivariable Cox proportional hazards regression was applied to predict risk factors for postoperative seizure recurrence within a 51-month follow-up period after PSM.

ELIGIBILITY:
Inclusion Criteria:

* 2 years old and above, no gender restriction, TSC gene monitoring with or without abnormality
* Diagnosis of tuberous sclerosis- related drug-resistant epilepsy
* Epilepsy course for more than 1 year
* Patients who have taken 3 or more reasonable choices with appropriate and tolerable antiepileptic drugs (excluding mTOR inhibitors and traditional Chinese medicine and prescriptions) had seizures more than 12 times in the 3 months before enrollment
* The family members agreed to enroll and signed the informed consent.

Exclusion Criteria：

* Obvious renal angiomyolipoma, pulmonary lymphoma leiomyomatosis, and subventricular giant cell astrocytoma
* Abnormal heart, lung, liver, and kidney functions and coagulation function
* Preoperative evaluation, it is considered that no surgical treatment is needed
* The patient received other craniocerebral surgical treatment within 1 year during the follow-up period

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from participating medical institutions
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
% of patients with ILAE grading | 3 years
  The grading made by ILAE for the classification of outcome with respect to epileptic seizures following epilepsy surgery. It contains a total of 6 levels. The higher the level, the worse the result. We will count the percentage of patients at each level.

SECONDARY OUTCOMES:
IQ | 3 years
  Wechsler Preschool and Primary Scale of Intelligence（WPPSI-III），Wechsler Intelligence Scale for Children (WISC-IV) and Wechsler Adult Intelligence Scale (WAIS-IV)，3 scales will be used for different ages to measure IQ. Higher scores mean better outcomes.
Quality of Life: QOLIE-31 | 3 years
  QOLIE-31 is suitable for patients 14 years and older. QOLCE-76 is applied to patients aged 2-13 by parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wei Z, Liu T, Cao D, Zhang K, Yang Z, Guo Q, Xu J, Liu S, Liu X, Guan Y, Peng Y, Yuan L, Chen L, Peng J, Han X, Chen C, Chen F, Lin W, Yu T, Zhao X, Wang J, Zhao R, Kuang S, Shi X, Zhai F, Zhang S, Feng W, Shan Y, Ding P, Qian R, Fang F, Chen S, Li H, Wang Y, Liu Q, Zhang H, Li W, Sun M, Zhang R, Liang S. Resective Surgery for Drug-Resistant Epilepsy in Patients With Tuberous Sclerosis Complex: A Prospective Nationwide Multicenter Cohort Study. Neurology. 2025 Nov 11;105(9):e214260. doi: 10.1212/WNL.0000000000214260. Epub 2025 Oct 16. PMID 41100778